CLINICAL TRIAL: NCT04154150
Title: Ketamine + Cognitive Training for Suicidality in the Medical Setting: Pilot
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Midway through this pilot study, funding was obtained to support a much larger study of the same interventions in this clinical population. Therefore the pilot study was halted so as not to compete with enrollment for the larger study.
Sponsor: Rebecca Price (Other)
Responsible Party: Sponsor-Investigator, Rebecca Price, Associate Professor of Psychiatry and Psychology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY19100041 (Part 1)
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Results first posted 2023-01-10 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Suicide, Attempted
MeSH Terms: conditions — Suicide, Attempted | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine + Cognitive Training (Experimental)
  Interventions: Drug: Intravenous ketamine; Behavioral: Cognitive training
- Ketamine + Sham Training (Sham Comparator)
  Interventions: Drug: Intravenous ketamine; Behavioral: Sham Training

INTERVENTIONS:
Drug: Intravenous ketamine — Single subanesthetic infusion of ketamine (0.5mg/kg)
Behavioral: Cognitive training — 8 sessions of computer-based cognitive training
  Arms: Ketamine + Cognitive Training
Behavioral: Sham Training — 8 sessions of computer-based sham training
  Arms: Ketamine + Sham Training

SUMMARY:
This project seeks to identify the acute and longer-term impact of a single dose of intravenous ketamine among suicidal patients referred for psychiatric consultation/liaison in the medical inpatient setting. The investigators will then test whether ketamine's rapid effects can be extended by introducing helpful information delivered by a computer-based training protocol. This work could ultimately lead to the ability to treat suicidality more efficiently and with broader dissemination by rapidly priming the brain for helpful forms of learning.

DETAILED DESCRIPTION:
NOTE: In the course of this pilot study, both the primary and secondary outcome measures were supplemented to provide additional, complementary information on the clinical effects of the study interventions, based on confirmation (through study team experience) of the feasibility of acquiring such additional information in the context of our study population, setting, and design.

ELIGIBILITY:
Inclusion Criteria:

Participants will:

1. be between the ages of 18 and 65 years
2. be a medical inpatient referred for psychiatric consultation/liaison due to suicidality
3. possess a level of judgment and understanding sufficient to agree to all procedures required by the protocol and must sign an informed consent document
4. be deemed an appropriate and reasonable medical candidate for intravenous ketamine by a physician authorized to prescribe medication to the patient during inpatient hospitalization

Exclusion Criteria:

1. Presence of current psychotic or autism spectrum disorder or current delirium
2. Use of a Monoamine Oxidase Inhibitor (MAOI) within the previous 2 weeks
3. Current pregnancy or breastfeeding
4. Reading level <5th grade as per WRAT-3 reading subtest
5. Past intolerance or hypersensitivity to ketamine
6. Patients taking any of the following medications: St John's Wort, theophylline, tramadol, metrizamide
7. Patients who have received ECT in the past 6 months prior to intake
8. Patients at risk for withdrawal related issues (e.g., delirium tremens, severe opiate withdrawal) or who present with substance-induced psychosis
9. Patients who, based on expressed preference and/or home geographic location, are deemed by the Psychiatric Consultation/Liaison service to be likely to receive inpatient psychiatric hospitalization at an alternate location outside of Western Psychiatric Institute & Clinic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.29 (14.80) | 35.44 (17.74) | 34.06 (16.06)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 2 | 5 | 7
  Female | 5 | 3 | 8
  Transgender (female-to-male) | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 5 | 8 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Montgomery Asberg Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] — depression severity; range 0-60; high score=worse outcome
  units on a scale | 39 (6.4) | 36.8 (6.3) | 37.8 (6.2)
Adult Suicide Ideation Questionnaire [Mean (Standard Deviation); unit: units on a scale] — suicidal ideation/thoughts; range 0-150; high score=worse outcome Population: Measure not acquired at baseline from 1 participant
  units on a scale
    number analyzed (Participants) | 6 | 9 | 15
    (all) | 85.0 (35.2) | 96.6 (31.5) | 91.9 (32.3)
Quick Inventory of Depressive Symptoms [Mean (Standard Deviation); unit: units on a scale] — Self-reported depression (range: 0-27; higher scores = worse outcome) Population: Measure not acquired at baseline from 2 participants
  units on a scale
    number analyzed (Participants) | 6 | 8 | 14
    (all) | 17.8 (3.1) | 14.4 (5.95) | 15.9 (5.1)
Scale for Suicide Ideation [Mean (Standard Deviation); unit: units on a scale] — suicidal ideation/thoughts; range 0-38; high score=worse outcome Population: Measure not acquired at baseline from 4 participants
  units on a scale
    number analyzed (Participants) | 4 | 8 | 12
    (all) | 30.3 (2.2) | 29.3 (1.7) | 29.6 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Rating Scale
Description: depression severity; range 0-60; high score=worse outcome
Time Frame: infusion +24 hours
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 7 | 9
score on a scale | 18.43 (8.5) | 15.44 (10.9)

2. Primary Outcome: Montgomery Asberg Depression Rating Scale
Description: depression severity; range 0-60; high score=worse outcome
Time Frame: infusion +5 days
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 7 | 8
score on a scale | 19.14 (9.8) | 16.13 (9.2)

3. Primary Outcome: Montgomery Asberg Depression Rating Scale
Description: depression severity; range 0-60; high score=worse outcome
Time Frame: infusion +12 days
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 3 | 7
score on a scale | 13.67 (14.2) | 17.29 (11.9)

4. Primary Outcome: Montgomery Asberg Depression Rating Scale
Description: depression severity; range 0-60; high score=worse outcome
Time Frame: infusion +1 month
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 3 | 6
score on a scale | 20.67 (7.6) | 14.00 (13.4)

5. Primary Outcome: Montgomery Asberg Depression Rating Scale
Description: depression severity; range 0-60; high score=worse outcome
Time Frame: infusion +3 months
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 4 | 7
score on a scale | 13.00 (13.6) | 14.71 (10.2)

6. Primary Outcome: Montgomery Asberg Depression Rating Scale
Description: depression severity; range 0-60; high score=worse outcome
Time Frame: infusion +6 months
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 5 | 7
score on a scale | 13.20 (14.7) | 17.43 (9.9)

7. Primary Outcome: Adult Suicide Ideation Questionnaire (Past Day Version)
Description: suicidal ideation/thoughts; range 0-150; high score=worse outcome
Time Frame: infusion +24 hours
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 6 | 9
score on a scale | 32.67 (8.45) | 41.89 (38.6)

8. Primary Outcome: Adult Suicide Ideation Questionnaire (Past Day Version)
Description: suicidal ideation/thoughts; range 0-150; high score=worse outcome
Time Frame: infusion +5 days
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 7 | 8
score on a scale | 20.00 (9.98) | 22.88 (10.7)

9. Primary Outcome: Adult Suicide Ideation Questionnaire (Past Day Version)
Description: suicidal ideation/thoughts; range 0-150; high score=worse outcome
Time Frame: infusion +12 days
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 6 | 7
score on a scale | 17.17 (13.4) | 31.86 (34.6)

10. Primary Outcome: Adult Suicide Ideation Questionnaire
Description: suicidal ideation/thoughts; range 0-150; high score=worse outcome
Time Frame: infusion +1 month
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 5 | 6
score on a scale | 23.60 (22.9) | 41.83 (48.0)

11. Primary Outcome: Adult Suicide Ideation Questionnaire
Description: suicidal ideation/thoughts; range 0-150; high score=worse outcome
Time Frame: infusion +3 months
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 5 | 6
score on a scale | 25.20 (26.2) | 37.50 (46.5)

12. Primary Outcome: Adult Suicide Ideation Questionnaire
Description: suicidal ideation/thoughts; range 0-150; high score=worse outcome
Time Frame: infusion +6 months
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 4 | 4
score on a scale | 29.5 (40.3) | 45.75 (60.9)

13. Secondary Outcome: Number of Participants With Occurrence of Suicidal Behaviors Per Medical Chart Review
Description: Number of participants with occurrence of any suicidal act (derived from medical chart) including: re-attempt, re-hospitalization for suicidality, or completed suicide
Time Frame: infusion +6 months
Population: All participants who were assigned to the arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 7 | 9
Participants | 3 | 4

14. Secondary Outcome: Number of Participants Reporting Suicidal Behaviors Per the Columbia Suicide Severity Rating Scale (CSSRS)
Description: Number of participants with occurrence of any suicidal act (derived from Columbia Suicide Severity Rating Scale interview; each of the following items was scored yes/no for the period since last assessment: re-attempt, re-hospitalization for suicidality, or completed suicide. Analyzed outcome measure is # of participants with 1 or more 'yes' responses.
Time Frame: infusion +6 months
Population: All participants who were assigned to the arm and were willing and able to complete at least one CSSRS interview at any point during follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 6 | 8
Participants | 1 | 1

15. Secondary Outcome: Quick Inventory of Depressive Symptoms
Description: Self-reported depression (range: 0-27; higher scores = worse outcome)
Time Frame: infusion +24 hours
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 6 | 9
score on a scale | 12.83 (4.1) | 11.22 (6.0)

16. Secondary Outcome: Quick Inventory of Depressive Symptoms
Description: Self-reported depression (range: 0-27; higher scores = worse outcome)
Time Frame: infusion +5 days
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 7 | 8
score on a scale | 9.86 (5.8) | 9.50 (6.9)

17. Secondary Outcome: Quick Inventory of Depressive Symptoms
Description: Self-reported depression (range: 0-27; higher scores = worse outcome)
Time Frame: infusion +12 days
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 6 | 7
score on a scale | 8.33 (7.1) | 9.86 (7.3)

18. Secondary Outcome: Quick Inventory of Depressive Symptoms
Description: Self-reported depression (range: 0-27; higher scores = worse outcome)
Time Frame: infusion +1 month
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 5 | 6
score on a scale | 9.60 (3.4) | 9.33 (7.0)

19. Secondary Outcome: Quick Inventory of Depressive Symptoms
Description: Self-reported depression (range: 0-27; higher scores = worse outcome)
Time Frame: infusion +3 months
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 5 | 6
score on a scale | 10.60 (7.1) | 9.17 (7.5)

20. Secondary Outcome: Quick Inventory of Depressive Symptoms
Description: Self-reported depression (range: 0-27; higher scores = worse outcome)
Time Frame: infusion +6 months
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 4 | 4
score on a scale | 10.00 (10.0) | 12.25 (10.6)

21. Secondary Outcome: Scale for Suicide Ideation
Description: suicidal ideation/thoughts; range 0-38; high score=worse outcome
Time Frame: infusion +24 hours
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure. Measure added to protocol after first 4 patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 2 | 5
score on a scale | 8.50 (12.0) | 0.80 (1.3)

22. Secondary Outcome: Scale for Suicide Ideation
Description: suicidal ideation/thoughts; range 0-38; high score=worse outcome
Time Frame: infusion +5 days
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 2 | 5
score on a scale | 0.50 (.71) | 6.60 (9.4)

23. Secondary Outcome: Scale for Suicide Ideation
Description: suicidal ideation/thoughts; range 0-38; high score=worse outcome
Time Frame: infusion +12 days
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 0 | 4
score on a scale |  | 4.50 (9.0)

24. Secondary Outcome: Scale for Suicide Ideation
Description: suicidal ideation/thoughts; range 0-38; high score=worse outcome
Time Frame: infusion +1 month
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 1 | 3
score on a scale | 13.00 | 4.67 (7.2)

25. Secondary Outcome: Scale for Suicide Ideation
Description: suicidal ideation/thoughts; range 0-38; high score=worse outcome
Time Frame: infusion +3 months
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 4 | 6
score on a scale | 4.00 (7.3) | 5.83 (9.2)

26. Secondary Outcome: Scale for Suicide Ideation
Description: suicidal ideation/thoughts; range 0-38; high score=worse outcome
Time Frame: infusion +6 months
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
Number analyzed (Participants) | 5 | 7
score on a scale | 5.40 (12.1) | 6.86 (9.2)

ADVERSE EVENTS:
Time Frame: 24 hours
Description: Adverse events were collected using the Patient Rated Inventory of Side Effects (PRISE; Rush et al 2004) instrument. Open-ended questions were also used to inquire about any additional adverse events not captured on the PRISE. Adverse events were tallied for all symptoms that were reported as new or worsening from pre-infusion baseline with onset during the infusion and/or within the subsequent 24hr period.
Arm/Group | Ketamine + Cognitive Training | Ketamine + Sham Training
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 7/7 | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine + Cognitive Training (N=7) | Ketamine + Sham Training (N=9)
anxiety (Psychiatric disorders) | 2 | 3
constipation (Gastrointestinal disorders) | 2 | 2
decreased energy (General disorders) | 1 | 2
diarrhea (Gastrointestinal disorders) | 0 | 1
difficulty sleeping: too little (Psychiatric disorders) | 3 | 3
difficulty sleeping: too much (Psychiatric disorders) | 0 | 1
dizziness (Nervous system disorders) | 2 | 2
dry mouth (Gastrointestinal disorders) | 1 | 1
emotional indifference (Psychiatric disorders) | 3 | 2
feeling 'high' (Nervous system disorders) | 1 | 0
headache (Nervous system disorders) | 2 | 3
increased appetite (Gastrointestinal disorders) | 1 | 2
loss of sexual desire (Reproductive system and breast disorders) | 0 | 1
nausea (Gastrointestinal disorders) | 3 | 0
restlessness (General disorders) | 1 | 2
sweating (General disorders) | 2 | 3
tremors (Nervous system disorders) | 0 | 1
trouble achieving orgasm (Reproductive system and breast disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Pilot study leading to small numbers of patients in each treatment arm. Descriptive statistics are reported without statistical analysis to directly compare groups, given the small number of patients within each group leading to low statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT04154150/Prot_SAP_000.pdf